CLINICAL TRIAL: NCT00309959
Title: A Phase II Evaluation of ABI-007 in the Treatment of Persistent or Recurrent Squamous or Nonsquamous Cell Carcinoma of the Cervix
Brief Title: ABI-007 in Treating Patients With Persistent or Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0127V; NCI-2009-00576 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0127V; CDR0000463520; GOG-0127V (Other: Gynecologic Oncology Group); GOG-0127V (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2014-12

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Small Cell Carcinoma; Cervical Squamous Cell Carcinoma; Recurrent Cervical Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Taxes; Albumin-Bound Paclitaxel

ARMS (1):
- Treatment (paclitaxel albumin-stabilized nanoparticle) (Experimental): Patients receive ABI-007 IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation — Given IV
  Other Names: ABI 007; ABI-007; Abraxane
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well ABI-007 works in treating patients with persistent or recurrent cervical cancer. Drugs used in chemotherapy, such as ABI-007, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Estimate the antitumor activity of ABI-007 in patients with persistent or recurrent squamous or nonsquamous cell carcinoma of the cervix who have failed on higher-priority treatment protocols.

II. Determine the nature and degree of toxicity of ABI-007 in this cohort of patients.

III. To determine the expression of the SPARC (secreted protein, acidic and rich in cysteine) protein in the tumor tissue and plasma (exploratory study) of patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study.

Patients receive ABI-007 IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and periodically during study for SPARC protein expression analysis by ELISA. Archived tumor tissue samples are also analyzed.

After completion of study treatment, patients are followed periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Persistent or recurrent squamous or nonsquamous cell carcinoma of the cervix with documented disease progression
* Histologic confirmation of the original primary tumor
* Measurable disease, defined as at least one target lesion that can be accurately measured in at least one dimension ≥ 20 mm when measured by conventional techniques, including palpation, plain x-ray, CT scan, or MRI, or ≥ 10 mm when measured by spiral CT scan

  * Tumors within a previously irradiated field will be designated as nontarget lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days after completion of radiotherapy
* Must have received 1 prior systemic chemotherapeutic regimen for management of advanced, metastatic, or recurrent squamous or nonsquamous cell carcinoma of the cervix

  * Chemotherapy administered as a radiosensitizer is not a systemic chemotherapy regimen
* Not eligible for a higher priority GOG protocol
* GOG performance status 0, 1, or 2
* No active infection requiring antibiotics
* Platelet count ≥ 100,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* SGOT and alkaline phosphatase ≤ 2.5 times ULN
* No neuropathy (sensory and motor) > grade 1
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No evidence of any other invasive malignancies within the past 3-5 years, except localized breast cancer, head and neck cancer, cervical cancer, or nonmelanoma skin cancer
* No pre-existing hearing loss/tinnitus > grade 1
* No concurrent amifostine or other protective agents
* Recovered from effects of prior surgery, radiotherapy, or chemotherapy
* Hormonal therapy directed at malignant tumor must be discontinued at least 1 week prior to study entry

  * Continuation of hormone replacement therapy permitted
* At least 3 weeks since prior biological therapy and immunotherapy
* No more than 1 prior cytotoxic chemotherapy regimen (either with single or combination cytotoxic drug therapy)

  * May have received 1 additional noncytotoxic (biologic or cytostatic) regimen, including monoclonal antibodies, cytokines, or small-molecule inhibitors of signal transduction
* No prior radiotherapy to any portion of the abdominal cavity or pelvis

  * Radiotherapy for the treatment of cervical cancer within the past 5 years allowed
  * Radiotherapy for localized breast cancer, head and neck or skin allowed provided completion > 3 years prior to study entry and remains free of recurrent or metastatic disease
* No prior chemotherapy for any abdominal or pelvic tumor

  * Chemotherapy for the treatment of cervical cancer within the past 5 years allowed
  * Prior adjuvant chemotherapy for localized breast cancer provided completion > 3 years prior to study entry and remains free of recurrent or metastatic disease
* No prior therapy with ABI-007 or any other taxane
* No prior anticancer treatment that would preclude study therapy
* No concurrent ritonavir, saquinavir, indinavir, nelfinavir, or anticonvulsants

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-11; Primary Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Alberts, Principal Investigator — Gynecologic Oncology Group
Locations (26):
- United States (26):
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Hospital Springfield, Springfield, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - Women's Cancer Care Associates LLC, Albany, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was opened to patient entry on November 6, 2006 and was closed to accrual on February 1, 2011.
Groups:
- ABI-007: ABI-007 125 mg/m2 IV weekly on day 1, 8, and 15 every 28 days (one cycle) until disease progression or adverse effects prohibit further therapy
Period: Overall Study
Arm/Group | ABI-007
Started | 37
Completed (Eligible and treated patients) | 35
Not Completed | 2
Not completed — Ineligible - no prior chemotherapy | 2

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | ABI-007
Number analyzed (Participants) | 35
Age, Customized [Number; unit: participants]
  <40 years | 6
  40-49 years | 15
  50-59 years | 10
  60-69 years | 3
  >70 yeats | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 30
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Objective Tumor Response Rate (Complete Response [CR] or Partial Response [PR]) Using RECIST Version 1.0
Description: RECIST 1.0 defines complete response as the disappearance of all target lesions and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Partial response is defined as at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of non-target lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required. In the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% decrease in the LD is required. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: CT scan or MRI if used to follow lesion for measurable disease every other cycle for the first 6 months; then every 3 months x 2; then every 6 months until disease progression for up to 5 years.
Population: Eligible and treated patients
Measure: Number; unit: participants
Arm/Group | ABI-007
Number analyzed (Participants) | 35
participants
  Partial response | 10
  Complete response | 0

2. Primary Outcome: Frequency and Severity of Observed Adverse Effects Assessed by Common Terminology Criteria for Adverse Events (CTCAE)
Time Frame: Up to 5 yearsAssessed every cycle while on treatment, 30 days after the last cycle of treatment, and up to 5 years in follow-up
Measure: Number; unit: participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1 (CTCAE v 3.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
- Grade 2 (CTCAE v 3.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
- Grade 3 (CTCAE v 3.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
- Grade 4 (CTCAE v 3.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
Arm/Group | Grade 0 | Grade 1 (CTCAE v 3.0) | Grade 2 (CTCAE v 3.0) | Grade 3 (CTCAE v 3.0) | Grade 4 (CTCAE v 3.0)
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35
participants
  Leukopenia | 11 | 10 | 12 | 3 | 0
  Thrombocytopenia | 30 | 4 | 0 | 1 | 0
  Neutropenia | 20 | 6 | 6 | 1 | 2
  Anemia | 3 | 6 | 22 | 4 | 0
  Nausea/Vomiting | 15 | 11 | 9 | 0 | 0
  Other gastrointestinal | 13 | 10 | 10 | 2 | 0
  Genitourinary | 34 | 1 | 0 | 0 | 0
  Neurotoxicity | 15 | 11 | 8 | 1 | 0
  Pain | 20 | 9 | 4 | 2 | 0
  Pulmonary | 31 | 1 | 2 | 2 | 0
  Cardiovascular | 34 | 0 | 1 | 0 | 0
  Fatigue | 8 | 7 | 15 | 5 | 0
  Metabolic | 24 | 5 | 2 | 4 | 0
  Dermatologic | 30 | 1 | 3 | 1 | 0
  Alopecia | 17 | 3 | 15 | 0 | 0
  Musculoskeletal | 32 | 2 | 1 | 0 | 0
  Auditory | 34 | 0 | 1 | 0 | 0
  Infection | 27 | 0 | 4 | 4 | 0
  SGOT | 34 | 1 | 0 | 0 | 0
  Alkaline phosphatase | 34 | 1 | 0 | 0 | 0
  Lymphatics | 31 | 2 | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment, and up to 5 years in follow-up
Arm/Group | ABI-007
Serious Adverse Events (participants affected / at risk) | 17/35
Other Adverse Events (participants affected / at risk) | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABI-007 (N=35)
Fever (General disorders) | 1
Death No Ctcae Term - Death Nos (General disorders) | 1
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Prolapse Of Stoma, Gi (Gastrointestinal disorders) | 1
Hemorrhage, Gi - Rectum (Vascular disorders) | 1
Infection with Normal Or Grade 1 Or 2 Absolute Neutrophil Count: Blood (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Wound (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 1
Edema: Limb (Blood and lymphatic system disorders) | 1
Creatinine (Metabolism and nutrition disorders) | 2
Gait/Walking (Musculoskeletal and connective tissue disorders) | 1
Neurology - Other (Nervous system disorders) | 1
Pain: Extremity-Limb (General disorders) | 1
Pain: Back (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Cystitis (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABI-007 (N=35)
Leukopenia (Blood and lymphatic system disorders) | 25
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 15
Anemia (Blood and lymphatic system disorders) | 32
Nausea/vomiting (Gastrointestinal disorders) | 20
Other gastrointestinal (Gastrointestinal disorders) | 22
GU (Renal and urinary disorders) | 1
Neurotoxicity (Nervous system disorders) | 20
Pain (General disorders) | 15
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 5
Cardiovascular (Cardiac disorders) | 1
Constitutional (Fatigue) (General disorders) | 27
Metabolic (Metabolism and nutrition disorders) | 11
Dermatologic (Skin and subcutaneous tissue disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 18
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 3
Auditory (Ear and labyrinth disorders) | 1
Infection (Infections and infestations) | 8
SGOT (Investigations) | 1
Alkaline phosphatase (Investigations) | 1
Lymphatics (Blood and lymphatic system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less